CLINICAL TRIAL: NCT05661331
Title: VIATORR Device Registry - Post-Market Clinical Follow-Up (PMCF) Registry of the GORE® VIATORR® TIPS Endoprosthesis With Controlled Expansion to Treat Portal Hypertension and Its Complications
Brief Title: VIATORR Device Registry
Status: Active, not recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VTR 21-09
Record Dates: First submitted 2022-11-29; First posted 2022-12-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ascites: N = Up to 88 treated patients and thereof, approximately 10 subjects with a pre-TIPS LVP frequency ≥ 2 LVP per month
  Interventions: Device: Transjugular intrahepatic portosystemic shunt
- Variceal bleeding: N = At least 88 treated patients and thereof, approximately 10 subjects enrolled with Child-Pugh class C
  Interventions: Device: Transjugular intrahepatic portosystemic shunt
- Other Primary Indication: Portal vein obstruction or thrombosis, pre-operative TIPS, hepatorenal Syndrome Type 1, hepatorenal Syndrome Type 2, other) N = Approximately 20 treated patients
  Interventions: Device: Transjugular intrahepatic portosystemic shunt

INTERVENTIONS:
Device: Transjugular intrahepatic portosystemic shunt — The GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion is indicated for use in the treatment of portal hypertension and its complications such as variceal bleeding and refractory ascites. The GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion is a current generation of the GORE® VIATORR® TIPS Endoprosthesis. The GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion was designed to build on the success of the GORE® VIATORR® TIPS Endoprosthesis. The GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion allows for intraoperative diameter control to reach a targeted portal pressure gradient.
  Other Names: TIPS

SUMMARY:
The primary objective is to confirm the clinical performance and safety of the GORE® VIATORR® TIPS (Transjugular Intrahepatic Portosystemic Shunt) Endoprosthesis with Controlled Expansion throughout the device functional lifetime of 3 years in real world setting.

The secondary objective is to collect information on quality of life after treatment with the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion.

Additionally, data will be collected on the safety and performance of the GORE TIPS Set when utilized.

DETAILED DESCRIPTION:
1. Registry Procedures

   1.1. Informed Consent Process All patients must provide informed consent prior to any registry related procedures. The original signed informed consent form will be retained in the subject records. A copy of the informed consent document will be given to the subject.

   1.1.1. Vulnerable Populations No vulnerable populations are included in this registry. 1.1.2. Emergent Cases Emergent cases, in which prior informed consent of the subject is not possible because of the subject's medical condition, can be enrolled in this registry by signing the inform consent before discharge.

   1.2. Enrollment The patient is considered enrolled when informed consent is obtained. 1.3. Screening All patients who sign an informed consent will be considered entered into the screening phase of the registry.

   The following evaluations will be conducted:
   * Informed consent
   * Inclusion / exclusion criteria
   * Demographics
   * Medical history including o Primary: variceal bleeding (gastric or esophageal), ascites (per EASL (European Association for the Study of the Liver) guidelines), other o Secondary: variceal bleeding, ascites (per EASL guidelines), hepatic hydrothorax, gastropathy, hepatorenal syndrome, other
   * Physical examination
   * Child-Pugh Score, MELD (Model for end-stage liver disease), MELD-Na (Model for end-stage liver disease including sodium level), Clif C AD (Acute Decompensation) Score.
   * Portal Hypertension details covering prior 12 months before ICF (Inform Consent Form) signature
   * HE (Hepatic Encephalopathy) Assessment
   * Medication
   * Alcohol intake
   * Pregnancy test
   * EQ-5D-5L (Health Questionnaire - 5 dimensions) Questionnaire
   * CLDQ (Chronic Liver Disease Questionnaire) Questionnaire 1.4. Screen Failure If the subject signed an informed consent and then is considered a screen failure prior to procedure, the Subject Identification (ID) will be entered into the Electronic Database Capture (EDC) system and the Inclusion / Exclusion Criteria Case Report Form (CRF) will be completed to reflect criteria not met. Additionally, the Completion / Discontinuation form has to be completed to capture when the subject is no longer enrolled in the registry.

   1.5. Procedure The GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion procedure will be performed according to standard practice of the enrolling institution and the IFU (Instructions for Use).

   No planned surgical concomitant procedures should be performed during the TIPS procedure. If any unplanned surgical concomitant procedures are required during the TIPS procedure the reason should be documented and entered into the Electronic Data Capture (EDC) system.

   The following details will be collected on the TIPS placement:

   • Access vein, starting vein and portal vein entry location
   * TIPS set used
   * Pre- and post-dilation details
   * Additional procedures performed
   * PSG (Portosystemic Gradient) measurements
   * Completion imaging (per site standard)
   * Adverse Events (as occurred) Any implanted GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion will be recorded on the subject's Procedure and Device Accountability electronic Case Report Forms (eCRFs). If a GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion was introduced into the vasculature and not implanted as part of the registry procedure (e.g., no shunt implant), the subject is considered an unsuccessful implant. The subject's Procedure, AE (Adverse Event), Device Accountability, and Device Deficiency eCRFs will be completed (as applicable), as well as a 30-day safety follow-up, where only AEs will be collected. After this 30-day safety follow-up, the Completion/Discontinuation form must be completed for patients with an unsuccessful GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion.

   Any procedural complications arising after enrollment of an eligible subject (signed ICF) will be treated per investigator's best medical judgment and recorded in the EDC system as an AE.

   1.6. HE Assessment Hepatic encephalopathy diagnosis detail should include covert and overt classification, history of recurrent HE prior to TIPS, HE diagnosis at time of TIPS, or HE at any time following TIPS procedure. Detail will be also collected on the HE medication therapy.

   1.7. Concomitant Medication Medication detail collected should include albumin, antibiotics, antivirals, alcohol dependence medication, antiplatelets/antithrombotics, chelating agents, corticosteroids, blood coagulation, diuretics, somatostatins, Proton Pump Inhibitors, laxatives, and beta-blockers.

   1.8. Imaging Images might be requested from sites for safety follow-up reasons. 1.9. Repeat Interventions Repeat interventions performed on the original pathology or directly on the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion following the initial treatment will be recorded in the EDC system. The underlying cause for repeat interventions should be recorded as an AE along with the treatment as specified.

   The following details will be collected on the TIPS revision:
   * Access vein, starting vein and portal vein entry location
   * TIPS set used
   * Pre- and post-dilation details
   * Additional procedures performed
   * PSG measurements
   * Completion imaging (per site standard)
   * Adverse Events (as occurred) If the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion is completely removed as part of the reintervention, then the subject is discontinued from the registry and should be followed as per the treating physician's standard of care.

   1.10. Follow Up The follow-up visits should be completed within an acceptable time frame and in accordance with the protocol-defined visit windows.

   Subjects will continue to be followed by the site's standard of care after completion of the registry.

   1.10.1. Discharge or Day 7 Visit The first visit after the procedure will be performed at discharge or day 7 post-surgery, whatever comes first.

   The following data will be collected during this visit:

   • Portal Hypertension - update on any new or existing portal hypertension symptoms and treatments since last visit

   • HE Assessment
   * Medication
   * TIPS imaging per site standard
   * Adverse Events

   1.10.2. FU (Follow-Up) Visit at 1, 3, 6, 12, 24 and 36 Months During the Follow-Up period, visits will be conducted per visit windows as listed above in Table 5.

   The following data will be collected during the follow-up visits:

   • Physical examination

   • Child-Pugh Score, MELD, MELD-Na, Clif C AD Score

   • Portal Hypertension - update on any new or existing portal hypertension symptoms and treatments since last visit

   • HE Assessment

   • Medication

   • EQ-5D-5L Questionnaire

   • CLDQ Questionnaire

   • TIPS imaging per site standard
   * Adverse Events (as occurred) 1.11. Subject Questionnaires Two health-related quality of life instruments will be used, EQ-5D-5L as a general instrument and CLDQ as disease-specific instrument (Chronic Liver Disease Questionnaire).

   1.12. Subject Withdrawal from the Registry A subject may withdraw from the registry at any time and should notify the investigator in this event. The investigator may also withdraw the subject from the registry at any time based on his / her medical judgment.

   If such withdrawal is due to problems related to the registry device safety or performance, the investigator shall ask for the subject's permission to follow his / her status / condition outside the clinical investigation.

   1.13. Subject Lost to Follow Up A subject will be considered lost to follow up and withdrawn from the registry once they have missed two consecutive follow-up visits and three documented attempts have been made by the investigator or designee to contact the subject or next of kin. One of the three documented attempts must include a certified letter. The subject's end date will be the last date of contact made with the subject.

   1.14. Subject Registry Completion A subject has completed the registry once the 36-month follow-up visit has been performed. Any subject that does not complete these requirements due to voluntary withdrawal, physician withdrawal, death, or any other reason will be considered a withdrawal. Subjects who miss two consecutive visits and three documented attempts will be considered lost to follow up. Subjects will not be provided with any medical care by the sponsor after registry completion or withdrawal.

   Subjects with a liver transplant or abandonment of the implanted device will exit the registry at that timepoint and no further follow-up information will be collected from these subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible for treatment with the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion for TIPS creation
2. Patient is ≥18 years of age
3. Capable of complying with protocol requirements, including follow-up
4. Signed informed consent by patient

Exclusion Criteria:

1. Unable or not willing to sign informed consent
2. Patient is enrolled in an investigational study
3. Patient has been previously enrolled in this registry
4. Pregnant or breastfeeding female at time of informed consent signature
5. Any other condition which in the judgement of the investigator would preclude adequate registry participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion for portal hypertension and its complications including, but not limited to, variceal bleeding and/or ascites.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Shunt primary patency through 3 years | Through 3 years
  Shunt primary patency is defined as freedom from reintervention due to shunt dysfunction (occlusion or thrombosis on imaging or significant stenosis confirmed by venography) or shunt occlusion. Intentional shunt occlusions of otherwise patent stents will not be considered a loss of primary patency.
  Shunt primary patency will be analyzed at 1, 3, 6, 12, 24 and 36 months. There is no formal hypothesis that will be tested for the primary endpoint. The analysis of the primary endpoint will be descriptive in nature.

SECONDARY OUTCOMES:
Technical success at day 0 | Day 0 - Intervention
  Successful delivery and deployment of the device to create or revise an intrahepatic shunt connection between the portal and hepatic circulations.
Reduction in PSG at day 0 | Day 0 - Intervention
  Difference between the pre-TIPS gradient (prior to TIPS device deployment) and the post-TIPS gradient (at completion of procedure).
Variceal rebleeding through 3 years | Through 3 years
  Variceal rebleeding is defined as any variceal bleeding event that occurs post procedure. The inability to control acute bleeding after device implant at time of procedure will count as a rebleeding event on day 0. Variceal rebleeding will be analyzed at 1, 3, 6, 12, 24 and 36 months.
Frequency of LVP (Large Volume Paracentesis) through 3 years | Through 3 years
  Any reported episode of LVP (> 5 L) following the TIPS procedure. LVP frequency will be analyzed at 1, 3, 6, 12, 24 and 36 months.
Quality of life (EQ-5D-5L) questionnaire compared to baseline at 1, 3, 6, 12, 24, 36 months | Through 3 years
  EQ-5D-5L questionnaire (With exception of France, refer to Section 5.13 in protocol). Each of the five dimensions comprising the The EQ-5D instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS). EQ-5D descriptive system is divided into five levels of perceived problems: LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems The EQ VAS scale goes from 0 to 100, with 100 meaning the best health possible
Quality of Life (CLDQ) questionnaire compared to baseline at 1, 3, 6, 12, 24, 36 months | Through 3 years
  CLDQ questionnaire (With exception of France, refer to Section 5.13 in protocol). The CLDQ is a short, easy to administer, produces both a summary score and domain scores, and correlates with the severity of liver disease. Higher score equates to worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jonel Trebicka, Prof Dr med, Principal Investigator — Universitätsklinikum Münster
Locations (7):
- Medical University of Vienna - Department of Internal Medicine III, Vienna, Austria
- Hôpital La Pitiè-Salpétrière, Paris, France
- Germany (2):
  - University Medical Center Freiburg, Department of Medicine II, Freiburg im Breisgau
  - Westfälische Wilhelms-Universität Münster, Münster
- Italy (2):
  - AOU Careggi, Florence
  - University Hospital Modena, Modena
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No